CLINICAL TRIAL: NCT06641700
Title: The Development and Prognosis of Gastric Cancer Based on Air Pollution and Metabolomics
Brief Title: Predictive Value of Air Pollution and Metabolomics for Gastric Cancer.
Status: Active, not recruiting | Type: Observational
Sponsor: Dong Peng (Other)
Responsible Party: Sponsor-Investigator, Dong Peng, Principal Investigator, First Affiliated Hospital of Chongqing Medical University
Organization: First Affiliated Hospital of Chongqing Medical University (Other)
Other Study IDs: 2024-221-02
Record Dates: First submitted 2024-10-13; First posted 2024-10-15 (Actual); Last update posted 2024-10-16 (Actual); Status verified 2024-10

CONDITIONS: Gastric Cancers
Keywords: gastric cancer; environment; air pollution; metabolomics; gut microorganisms
MeSH Terms: conditions — Stomach Neoplasms | interventions — Diagnosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- the gastric cancer group: Pre-operative gastric cancer diagnosed by pathological biopsy in our clinic.
  Interventions: Diagnostic Test: diagnosed with gastric cancer
- the contol group: Adults with no history of malignancy and willing to participate in this study.

INTERVENTIONS:
Diagnostic Test: diagnosed with gastric cancer — Pathological biopsy confirmed the diagnosis of gastric cancer.
  Groups: the gastric cancer group

SUMMARY:
As one of the common malignant tumours worldwide, gastric cancer continues to have a high incidence and mortality rate, especially in Asia. Although a large number of studies have focused on its underlying genetic and lifestyle factors, the specific role of environmental factors in gastric cancer development and progression has not been fully elucidated. Air pollution, a growing environmental problem, and its major components such as PM2.5, PM10, and NO2 have been shown to be closely associated with the occurrence and development of many chronic diseases. Recent studies have gradually revealed the association between air pollution and certain cancer types (e.g., lung cancer), but its relationship with gastric cancer remains relatively unexplored. Against this background, the application of metabolomics provides new perspectives and methods to study the association between gastric cancer and environmental factors. Metabolomics is capable of systematically analysing the metabolite composition and changes in individuals under different environmental exposures, revealing the potential effects of environmental factors, such as air pollution, on individual metabolic functions. By combining air pollution data and metabolomics analysis, investigators can deeply explore the role of environmental factors in the occurrence, development and prognosis of gastric cancer, and thus provide a scientific basis for the development of prevention and treatment strategies.

DETAILED DESCRIPTION:
In this study, clinical data, blood, urine and stool specimens were collected by including patients in the healthy control group and gastric cancer group. The air pollution indicators, metabolomics determination and macro genomic determination were extracted from clinical data, blood and stool respectively. The extracted air pollution, metabolomics and intestinal microbiota data were integrated and analysed. Based on machine learning, a comprehensive model was constructed to screen the key indicators that play a role in the development of gastric cancer and construct a prediction model for gastric cancer development. The aim of this study is to investigate how environmental, metabolic and microbiota factors affect the occurrence and development of gastric cancer. Secondly, metabolic markers specific to gastric cancer patients can also be identified, providing a basis for early diagnosis, early intervention and individualised treatment.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of gastric cancer confirmed by pathology or cytology;
* aged >18 years;
* not received chemotherapy, radiotherapy, targeted therapy or immunotherapy;
* post-operative pathological stages other than stage IV, or no liver, lung or other organs as confirmed by CT, MRI, B-ultrasound imaging.

Exclusion Criteria:

* Patients with systemic diseases such as severe cardiorespiratory insufficiency affecting the choice of treatment regimen;
* inappropriate for enrolment as assessed by the investigator;
* incomplete clinical data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All adult patients diagnosed with gastric and undergoing radical surgery for gastric cancer at the study centre may be included in the gastric cancer group.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2024-10-01 (Actual); Primary Completion 2026-10-01 (Estimated); Study Completion 2029-10-01 (Estimated)

PRIMARY OUTCOMES:
Rate of postoperative complications | From date of surgery until the date of first documented postoperative complication, assessed up to 2 months after surgery.
  Surgical complications was defined as any postoperative complication occurring during the postoperative hospitalisation period.

SECONDARY OUTCOMES:
Overall survival | From date of diagnosis until the date of death from any cause or or loss to follow-up, whichever came first, assessed up to 60 months
  Overall survival was defined as time from date of diagnosis until the date of death from any cause or or loss to follow-up.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Chongqing Medical University, Chongqing, Chongqing Municipality, China

IPD SHARING:
Plan to Share IPD: No